



## Antimicrobial Stewardship Program Based on the Detection and Monitoring of Patients with Clostridium difficile infection.

NCT02951481 Protocol ID: JMA-MET-2016-01

Version 2.0 February 15, 2016

Infectious Diseases Unit. Fundación de Investigación "i+12" University Hospital "12 de Octubre"





## Patient Information Sheet.

You (or your relative) have been diagnosed with *Clostridium difficile* infection. This microorganism is responsible for most cases of **diarrhea associated with antibiotic treatment**, especially among hospitalized patients. Antibiotic treatment alters the normal intestinal flora and facilitates the overgrowth of this bacterium.

The symptoms are diarrhea, with or without abdominal pain and fever. Typically, the disease is cured in a few days with proper treatment, although there may be **a small percentage** of patients who develop a **severe infection** due to important inflammation of the colon.

In addition, a **20-30% of patients** diagnosed with a *Clostridium difficile* infection may have a **recurrence** and develop diarrhea again in the following months beyond the end of treatment, especially if they have to receive a new antibiotic treatment for some other reason.

Clostridium difficile produces spores that are found in the stools of infected patients. These spores are very resistant and, if hygiene measures are not optimal, they can remain on your skin and on the surfaces that you touch. While you still suffer from diarrhea, you can eliminate these spores through your stools.

Health workers can spread the spores and transmit the bacteria to other patients after treating you, that's why **contact precautions** have to be established. These measures include isolation in a single room, which you shouldn't leave unless it is necessary, and the use of gloves and gowns by health workers and your relatives while they are in the room, followed by hand washing with soap and water once they go out of the room.

**Don't be alarmed**, it's not common that healthy individuals develop the disease in the absence of antibiotic treatment and, on the other hand, transmission is easily avoided if **proper hygiene measures** are taken. The spores are removed with **soap and water**, so it is important for you and your relatives to wash your hands frequently, especially after using the bathroom and before touching or preparing food.

While you continue with diarrhea you should avoid using the same toilet as other family members. In addition, toilet bowl, the device flush, toilets and kitchen countertops should be cleaned with a mixture of bleach and water (1 part bleach to 10 parts water).

With our program we will provide you a closer medical monitoring both during admission and after discharge, by telephone contact or in person in the outpatient's clinic, if necessary, up to 8 weeks after the end of treatment for the *C. difficile* infection.

The University Hospital 12 de Octubre Ethics Committee has approved this project and all the information related to the study will be strictly confidential and treated according to the Organic Law 15/1999 on Protection of Personal Data.



## **Informed consent**

The intention of our project is to improve treatment and monitoring of patients with *Clostridium difficile* infection in our hospital.

As patient infected by this microorganism, we offer you the opportunity to participate in this study. For you, it would involve a closer monitoring by an Infectious Diseases physician while you are hospitalized. Once you are discharged, you will be contact weekly by phone or by email for 8 weeks after the end of treatment.

By this telephone calls, we will ensure that symptoms of *Clostridium difficile* infection do not recur. Besides, a phone number will be provided for you to call during working days in case of new symptoms, indication of antibiotic treatment for another reason or need for consultation.

Your clinical data will be collected and subsequently analyzed anonymously to know the benefits of our intervention.

**Study title:** "Antimicrobial Stewardship Program Based on the Detection and Monitoring of Patients with *Clostridium difficile* infection".

| my legal representative (name) | declare that |
|---|---|
| I read the information that the investigator has given me. | |
| I had the opportunity of asking any question about the study. | |
| I talked to Dr / Dr | |
| I understand that my participation is voluntary. | |
| I understand that I can leave the study: | |
| <ol> <li>Whenever I want.</li> <li>Without the need for giving any explanation.</li> </ol> | |
| 3. Without any influence on my regular medical care. | |

Date and signature of the patient (Or legal representative)

I consent freely to participate in the study

Date and signature of the investigator